CLINICAL TRIAL: NCT03431727
Title: Sleep Apnea, Circulation and Metabolism in Acromegaly - Before and After Treatment
Brief Title: Acromegaly - Before and After Treatment
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: 1-10-72-126-16
Record Dates: First submitted 2017-12-22; First posted 2018-02-13 (Actual); Last update posted 2020-12-07 (Actual); Status verified 2020-12

CONDITIONS: Acromegaly; Growth Hormone Treatment; Sleep Apnea; Cardiovascular Diseases; Bone Diseases
MeSH Terms: conditions — Acromegaly; Sleep Apnea Syndromes; Cardiovascular Diseases; Bone Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples and tissue will be kept in a locked freezer thorughout the study period
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to investigate sleep apnea, circulation and metabolism in acromegaly before and after surgery and/or medical treatment.

DETAILED DESCRIPTION:
Acromegaly is a rare disease caused by a growth hormone (GH) producing pituitary adenoma. Surgery is primary treatment, whereas medical treatment with a somatostatin analogue (SA), which suppresses GH secretion and reduces tumour size, is used when surgery is insufficient or unfeasible. Acromegaly is associated with metabolic abnormalities which contributes to an increased morbidity and mortality if left untreated. To which extend these abnormalities reverses after treatment, and if treatment modality influences the outcome, remain elusive. The aim of the study is to investigate sleep apnea, circulation and metabolism in acromegaly before and after surgery and/or medical treatment

ELIGIBILITY:
Inclusion Criteria:

* Recently diagnosed with acromegaly
* Age above 18
* Written consent

Exclusion Criteria:

- Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Newly diagnosed acromegalic patients
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2017-10-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Sleep apnea | At baseline (time of diagnosis) and at an average of 1 years treatment
  ApneaLinkAir: respiratory effort, puls, oxygen saturation, nasal flow and snoring
Circulation | At baseline (time of diagnosis) and at an average of 1 years treatment
  Sphygmocor: central arterial pressure and pulse wave velocity
Bone metabolism | At baseline (time of diagnosis) and at an average of 1 years treatment
  HRpQCT scan

SECONDARY OUTCOMES:
Heartfunction | At baseline (time of diagnosis) and at an average of 1 years treatment
  Echocardiography
Substrate metabolism; signaling proteins | At baseline (time of diagnosis) and at an average of 1 years treatment
  Western blotting
Substrate metabolism; gene targets | At baseline (time of diagnosis) and at an average of 1 years treatment
  qPCR
Energy expenditure | At baseline (time of diagnosis) and at an average of 1 years treatment
  Indirect calorimetry
Body composition | At baseline (time of diagnosis) and at an average of 1 years treatment
  DXA scan
Physical activity | At baseline (time of diagnosis) and at an average of 1 years treatment
  Sensoriband

CONTACTS AND LOCATIONS:
Overall Officials: Jens Otto L Jørgensen, Porfessor, Principal Investigator — Aarhus University Hospital, Department of internal medicine and endocrinology
Locations (1):
- Aarhus University Hospital, Department of internal medicine and endocrinologi, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No